CLINICAL TRIAL: NCT01823302
Title: Effect of a New Growing-up Milk on Growth and Nutrient Adequacy in Children With Picky-eating Behaviors
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 9601A1-4000
Record Dates: First submitted 2013-03-21; First posted 2013-04-04 (Estimated); Last update posted 2013-04-04 (Estimated); Status verified 2013-03

CONDITIONS: Picky Eating Behaviors
Keywords: Children with picky-eating behaviors; Children aged 2.5 - 5 years; reported by caregivers; with weight-for-height z-scores ≤ 25th percentile at enrollment
MeSH Terms: interventions — Nutrition Assessment

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- nutritional counseling (Other): nutritional counseling
  Interventions: Other: nutritional counseling
- nutritional counseling and milk-based supplement (Other): nutritional counseling plus oral milk-based nutrition supplement
  Interventions: Dietary Supplement: nutrition counseling plus oral milk-based nutritional supplement

INTERVENTIONS:
Dietary Supplement: nutrition counseling plus oral milk-based nutritional supplement — Study group subjects were instructed to consume at least 2 servings (230 mL per serving) of an oral milk-based nutritional supplement daily, in addition to their regular diet, for a total of 120 (±3) days.
  Arms: nutritional counseling and milk-based supplement
Other: nutritional counseling — nutritional counseling
  Arms: nutritional counseling

SUMMARY:
The primary objective of the study was to compare the change in z-scores for growth during a 120-day study period in children with picky eating behaviors who were randomly assigned to receive nutrition counseling only (control group) or nutrition counseling plus an oral milk-based nutritional supplement (study group). The secondary objectives of the study were to compare the following between the control and study groups: a) dietary macro- and micro-nutrient intakes; b) quantitative ultrasound bone measurements of radius and tibia; and c) incidence of common illnesses (diarrhea, upper and lower respiratory tract). The safety objective of the study was to compare the frequency of adverse events (AE) among the control group and study group subjects.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 30-60 months with PE behavior as reported by caregivers and whose weight-for-height was ≤25th percentile according to World Health Organization (WHO) Child Growth Standards were eligible for inclusion.

Exclusion Criteria:

* Current acute or chronic illness, food allergies, lactose intolerance, dietary restrictions precluding dairy foods, any genetic disorder that may compromise growth and/or food intake, cognitive or developmental disorders, or medications that may influence study outcomes.

Ages: 30 Months to 60 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 165 (Actual)
Dates: Start 2010-02; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Effect of a new growing-up milk on growth and nutrient adequacy in children with picky-eating behaviors | baseline to Day 120, as well as from baseline to Days 30, 60 and 90, and over the entire study period based on repeated measures analysis.
  The primary efficacy evaluation was growth, including the change in weight-for-height z-score from baseline to Day 120, as well as from baseline to Days 30, 60 and 90, and over the entire study period based on repeated measures analysis.

SECONDARY OUTCOMES:
Effect of a new growing-up milk on growth and nutrient adequacy in children with picky-eating behaviors | baseline to Day 120, as well as from baseline to Days 30, 60 and 90, and over the entire study period based on repeated measures analysis.
  Secondary efficacy evaluations included: dietary macro- and micro-nutrient intakes, quantitative ultrasound measurements of the radius and tibia, and incidence of common illnesses (diarrhea, and upper and lower respiratory tract infection).

OTHER OUTCOMES:
Effect of a new growing-up milk on growth and nutrient adequacy in children with picky-eating behaviors | baseline to Day 120, as well as from baseline to Days 30, 60 and 90, and over the entire study period based on repeated measures analysis.
  Safety was evaluated through the recording and monitoring of adverse events.
•Effect of a new growing-up milk on growth and nutrient adequacy in children with picky-eating behaviors | baseline to Day 120, as well as from baseline to Days 30, 60 and 90, and over the entire study period based on repeated measures analysis
  dietary macro- and micro-nutrient intakes
•Effect of a new growing-up milk on growth and nutrient adequacy in children with picky-eating behaviors | baseline to Day 120, as well as from baseline to Days 30, 60 and 90, and over the entire study period based on repeated measures analysis
  quantitative ultrasound measurements of the radius and tibia
•Effect of a new growing-up milk on growth and nutrient adequacy in children with picky-eating behaviors | baseline to Day 120, as well as from baseline to Days 30, 60 and 90, and over the entire study period based on repeated measures analysis
  and incidence of common illnesses (diarrhea, and upper and lower respiratory tract infection).

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoyang Sheng, Professor, Principal Investigator — Xinhua Hospital Affiliated to Shanghai Jiaotong
Locations (2):
- China (2):
  - Xinhua Hospital Affiliated to Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Xinhua Hospital Affiliated to Shanghai Jiaotong, Shanghai, Shanghai Municipality